CLINICAL TRIAL: NCT04660682
Title: A Comparison of the Long Term Effects of the Traditional and Modified Posterior Shoulder Stretching Exercise on Shoulder Mobility, Pain, Ultrasonographic Parameters, Proprioception, Strength, Functionality, and Disability Level in Subacromial Impingement Syndrome
Brief Title: A Comparison of the Long Term Effects of the Traditional and Modified Posterior Shoulder Stretching Exercise in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Halime Ezgi TÜRKSAN, MSc, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3032-GOA
Record Dates: First submitted 2020-11-28; First posted 2020-12-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Glenohumeral Internal Rotation Deficit, Modified Cross-body Stretching
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: There are 3 groups. The first group will receive the modified static cross-body posterior shoulder stretching and the standard physiotherapy program. The second group will receive traditional static cross-body posterior shoulder stretching and the standard physiotherapy program. The Control group will receive sham stretching and the standard physiotherapy program. In standard physiotherapy program, there are TENS, hot-pack, posture, proprioceptive, and strengthening training. The treatment program will last for eight weeks. Patients will receive the treatment program 5 days a week under the physiotherapist's supervision and 2 days a week as a home program.
Who Masked: Participant
Masking Description: All of the participants must have subacromial impingement syndrome with glenohumeral internal rotation deficit (Bilateral IRROM difference ≥ 15º )
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Modified static cross-body posterior shoulder stretching group (Experimental): The participants will perform active-assistive static stretching in the modified cross-body stretching position. Additionally, they will receive standard physiotherapy program.
  Interventions: Other: Modified static cross-body posterior shoulder stretching
- Traditional static cross-body posterior shoulder stretching group (Experimental): The participants will perform active-assistive static stretching in the traditional standing cross-body stretching position. Additionally, they will receive standard physiotherapy program.
  Interventions: Other: Traditional static cross-body posterior shoulder stretching
- Control Group (Active Comparator): The participants in this group will receive sham stretching and standard physiotherapy.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Modified static cross-body posterior shoulder stretching — For the modified cross-body position patient will be positioned in the side-lying position to limit the scapular abduction, and the patient aligned his/her forearms to limit the ER of the humerus while moving into horizontal adduction (HAdd). First, we will ask the patient to pull his/her arm into HAdd to the physiological barrier of the ROM, and then the patient will perform active-assistive static stretching with the help of the other hand for 30 seconds. The stretching will perform five repetitions with 10-sec rest between stretches. Each stretching will begin from a new physiological barrier of the HAdd ROM. Patients will also receive the standard physiotherapy program consists of physical agents, posture, proprioceptive, and strengthening exercises. The treatment program will be performed 5 days a week under the physiotherapist's supervision and 2 days a week as a home program for 8 weeks.
  Arms: Modified static cross-body posterior shoulder stretching group
Other: Traditional static cross-body posterior shoulder stretching — For the traditional static cross-body posterior shoulder stretching, in the standing position, the patient will perform cross-body stretch alone by active-assistive pulling the humerus across the body into HAdd with the opposite arm, without concern for scapular stabilization for 30 sec. The stretching will perform five repetitions with 10-sec rest between stretches. Each stretching will begin from a new physiological barrier of the HAdd ROM. Patients will also receive the standard physiotherapy program consists of physical agents, posture, proprioceptive, and strengthening exercises. The treatment program will be performed 5 days a week under the physiotherapist's supervision and 2 days a week as a home program for 8 weeks.
  Arms: Traditional static cross-body posterior shoulder stretching group
Other: Control Group — In sham stretching, the patient will be positioned in the traditional static cross body posterior shoulder stretching position, and then the patient will perform active-assistive HAdd ROM without enough stretching of the relevant tissue. Active assistive ROM will be stopped before reaching the individual PST measurement result (in this way, sham stretching will be performed without proper stretching of the relevant tissue). The HAdd ROM exercise will be performed 5 times. Patients will also receive the standard physiotherapy program consists of physical agents, posture, proprioceptive, and strengthening exercises. The treatment program will be performed 5 days a week under the physiotherapist's supervision and 2 days a week as a home program for 8 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate and compare the long term effects of traditional and modified static cross-body posterior shoulder stretching training in individuals with subacromial impingement syndrome (SIS) having glenohumeral internal rotation deficit (GIRD). Modified cross body posterior shoulder stretching group will receive static stretching in the modified cross-body stretching position and standard physiotherapy program. The traditional cross body posterior shoulder stretching group will receive static stretching and standard physiotherapy program. The Control group will receive only sham stretching and standard physiotherapy program.

DETAILED DESCRIPTION:
SIS is the most common cause of pain and shoulder dysfunction. The etiology of SIS depends on many factors including tightness of the posterior shoulder structures. Posterior shoulder tightness (PST) narrows the subacromial space and forces anterior-superior migration of the humeral head over the glenoid fossa and, it could cause limitation of the internal rotation (IR) and horizontal adduction range of motion (ROM). GIRD is known as loss of IR ROM in the glenohumeral joint. In the SIS, limitation IR ROM has been reported. Supraspinatus tendon thickness can change, subacromial space may become narrower and joint position sense (JPS) could be decreased in SIS patients. The effectiveness of traditional static cross body posterior shoulder stretching on various parameters such as shoulder rotational ROM or pain was studied and proved in the literature. Traditional static cross body posterior shoulder stretching could reduce subacromial symptoms and improve shoulder ROM with some disadvantages such as inadequate control of the scapula and glenohumeral rotation. To prevent accessory abduction of the scapula, restrict the external rotation ROM of the humerus and provide isolated posterior capsule stretching, Wilk et al. (2013) recommend the use of modified cross-body stretching for IR ROM increase. In the modified cross-body position, the patient is positioned in a more advantageous way. In the literature, although modified cross-body posterior stretching seems effective on SIS symptoms there is no research about the comparison of the long-term effects of the traditional and modified static cross-body posterior shoulder stretching exercises in individuals with SIS having GIRD. Therefore, whether modified stretching is superior to traditional stretching is not known. Our study aims to investigate and compare the long term effects of the traditional static cross-body posterior shoulder stretching exercise and modified static cross-body posterior shoulder stretching exercise in individuals with SIS having GIRD on shoulder IR ROM, GIRD, PST, pain, external rotation ROM, JPS, subacromial space, supraspinatus tendon thickness, posterior capsule thickness, the occupational ratio of the supraspinatus tendon in the subacromial space, muscle strength and shoulder function and disability level. Stretching groups will receive either traditional or modified static cross-body posterior shoulder stretching exercise and standard physiotherapy program. The Control group will receive only sham stretching and standard physiotherapy program. Standard physiotherapy program consists of electrotherapy, posture, proprioceptive, and strengthening exercises. The treatment program will be performed 5 days a week under the physiotherapist's supervision and 2 days a week as a home program for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome
* Glenohumeral internal rotation range of motion of the affected shoulder should be less than other shoulder and bilateral shoulder internal rotation range of motion difference should be ≥15 º
* Pain with resisted arm elevation or external rotation as well as a minimum of 3 of 5 positive subacromial impingement syndrome tests, painful arc, pain or weakness with resisted external rotation, Neer, Hawkins and Jobe tests .
* Ability to complete the entire study procedure

Exclusion Criteria:

* A 50% limitation of passive shoulder range of motion in >2 planes of motion
* Pain >7/10
* A history of fracture to the shoulder girdle
* Systemic musculoskeletal disease
* History of shoulder surgery,
* Glenohumeral instability (positive apprehension, relocation or positive sulcus test) or positive findings for a full thickness rotator cuff tear (positive lag sign, positive drop arm test, or marked weakness with shoulder external rotation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of shoulder internal rotation range of motion (with bubble inclinometer)
Glenohumeral internal rotation deficit | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of glenohumeral internal rotation deficit (with bubble inclinometer)

SECONDARY OUTCOMES:
Posterior shoulder tightness | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of posterior shoulder tightness (with bubble inclinometer)
Pain intensity | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of visual analog scale score in activity and rest
Joint position sense | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of shoulder joint repositioning angle errors for external rotation 0-45 degree, for internal rotation 0-45 degree, for scapular plane elevation 0-100 degree (with bubble inclinometer)
Isometric strength | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of shoulder abduction, internal rotation, and external rotation isometric strength (in kg, with hand held dynamometer)
Subacromial space | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of subacromial space at neutral (0 degree), 30, 45, and 60-degree scapular plane elevation(with Ultrasound)
Supraspinatus tendon thickness | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of supraspinatus tendon thickness (with Ultrasound)
Shoulder external rotation range of motion | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of shoulder external rotation range of motion (with bubble inclinometer)
Posterior capsule thickness | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of posterior capsule thickness (with Ultrasound)
Occupational ratio of the supraspinatus tendon in the acromial-humeral space | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of occupational rate of the supraspinatus tendon in the acromial-humeral space
Shoulder Function | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of Modified Constant-Murley Score
Upper extremity function | Baseline, 8 weeks, 12 weeks, 24 weeks
  Change of disabilities of the arm, shoulder, and hand (DASH) score

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, PT, Study Director — Dokuz Eylul University Physical Therapy and Rehabilitation Department; Mehmet ERDURAN, MD, Study Director — Dokuz Eylul University; Onur BAŞÇI, MD, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University Physical Therapy and Rehabilitation Department, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No